CLINICAL TRIAL: NCT01901926
Title: Impact of Non Surgical Periodontal Treatment on Glycemic Control in Type II Diabetics
Brief Title: Periodontal Treatment and Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Salman Aziz, Senior Post Graduate Resident (Dentistry), Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Salman-0509
Record Dates: First submitted 2013-06-12; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodontal Treatment (Active Comparator): Periodontal Treatment in the form of Full mouth scaling and root planning will be given at one time only i.e. at baseline after full mouth dental checkup.
  Checkup will be repeated at 3, 6 & 9 month interval along with HbA1C levels
  Interventions: Procedure: Non Surgical Periodontal Treatment
- Non treatment group (No Intervention): this group will only receive detailed dental check ups at the specified time 0, 3, 6 and 9 months respectively and there will be no scaling done. HbA1C levels will be estimated at the above specified times

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment — one time intervention in the form of scaling and root planing
  Arms: Periodontal Treatment

SUMMARY:
The purpose of this study is to determine the effects of non surgical periodontal treatment on glycemic control in type II diabetics.

DETAILED DESCRIPTION:
The selected patients in treatment group will be given mechanical periodontal treatment in the form of scaling and root planning while the non intervention group patients will not receive treatment until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of Type 2 Diabetes Mellitus for at least 2 years
* HbA1C values >6.5 % as per ADA criteria
* non smokers
* Patients with at least 16 standing teeth
* At least 8 teeth with one site having Mild to Moderate periodontal disease

Exclusion Criteria:

* Smokers
* Type 2 Diabetics with complications e.g. renal, ophthalmic etc
* Patients with chronic infections
* Patients who get hospitalized or have to change their medications during the course of study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C levels from base line at 3, 6 and 9 months | 3 months, 6 months, 9 months
  HbA1C levels will be recorded and any change in percentage noted

SECONDARY OUTCOMES:
Bleeding on Probing | Base Line, 3 months, 6 months and 9 months
  a change in the above mentioned periodontal parameters will be recorded at the specified times Bleeding on probing will be recorded as Yes or No for each tooth
Clinical Attachment Loss | Base Line, 3 months, 6 months, 9 months
  A change in the above mentioned periodontal parameter will be recorded at the specified times Clinical Attachment loss will be recorded in millimeters for each tooth
Periodontal Pocket Depth | Base Line, 3 months, 6 months, 9 months
  A change in Periodontal pocket will be measured in millimeters for the above mentioned time frame

OTHER OUTCOMES:
Fasting Blood Glucose | Base Line, 3, 6 and 9 Months
C-Reactive Protein | Base Line, 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Salman Aziz, FCPS, MFDS, Principal Investigator — Pakistan Institute of Medical Sciences
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Federal Capital, Pakistan